CLINICAL TRIAL: NCT03053024
Title: An Observational Study of Bortezomib (BTZ) Treatment on Mantle Cell Lymphoma (MCL) in China
Brief Title: Study of Bortezomib (BTZ) Treatment on Mantle Cell Lymphoma (MCL) in Chinese Participants
Status: Completed | Type: Observational
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108287; 26866138MCL4001 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Lymphoma, Mantle-Cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Relapse/refractory MCL (rrMCL ) Participants: Participants characteristics and treatment pattern of relapsed/refractory mantel cell lymphoma [rrMCL]) participants treated by Bortezomib (BTZ) will be observed for cohort 1.
- Cohort 2: Newly Diagnosed MCL Participants: Participants characteristics and treatment pattern of newly diagnosed MCL participants (if more than 20% of total BTZ-treated MCL) will be analysed for cohort 2.

SUMMARY:
The purpose of the study (retrospective and prospective) is to describe participant and disease characteristics and treatment pattern of Bortezomib treated mantle cell lymphoma (MCL) participants in China.

ELIGIBILITY:
Inclusion Criteria:

* Participants that have been hospitalized for MCL after January 1st 2009.
* Biopsy proven MCL as evidenced by histology with either immunohistochemistry (IHC) or t(11,14) translocation
* Retrospective group: Participants who have finished BTZ treatment before the study initiation as judged by participating site physician
* If participant isn't accessible for oral or written informed consent, ICF can be waived after approved by the IRB
* Prospective group: Participants who are on BTZ at the time of study initiation or start BTZ after study initiation

Exclusion Criteria:

* Participants with documented diagnosis of other cancers prior to or at the presence of the diagnosis of MCL
* Participants enrolled in interventional clinical trials of BTZ or any other drug for MCL
* Prospective group: Participants with contraindication listed in the prescribing information of BTZ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study include mantle cell lymphoma (MCL) participants who were or will be treated by Bortezomib (BTZ) per routine clinical care in multiple tertiary care hospitals after January 1st 2009. Both newly diagnosed MCL participants and relapsed/refractory MCL participants will be included.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Demographic Characteristic of Participants in Prospective Group: Age | Baseline
  Continuous variable (age) will be summarized using descriptive statistics.
Participants Disease Status (newly diagnosed MCL or relapsed/refractory mantel cell lymphoma [rrMCL]) Treated With BTZ | Baseline
  Categorical variable (disease status) will be summarized using a frequency distribution with the number and percentage of participants in each category. Treatment response will be analyzed by this variable if newly diagnosed MCL patients account for more than 20 percent (%) of total.
Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline
  A worsening in Eastern Cooperative Oncology Group (ECOG) performance status score was defined as greater than or equal to 1-point increase from Baseline. ECOG is a 5-point scale 0=Fully active, 1=Ambulatory, carry out work of sedentary nature, 2=Ambulatory, capable of all self-care, 3=Capable of limited self-care, confined to bed or chair more than 50% of waking hours, 4=Completely disabled, no self-care, totally confined to bed or chair, 5=Dead.
Ann Arbor Stage | Up to Follow-up (approximately 22 months)
  Ann Arbor stage can be obtained from imaging results or directly from admission records. Ann Arbor stage describes areas of involvement; Stage I(IE) - One lymph node region or extralymphatic site (IE); Stage II(IIE)- Two or more lymph node regions or at least one lymph node region plus a single localized extralymphatic site (IIE) on the same side of the diaphragm; stage III (IIIE, IIIS)-Lymph node regions or lymphoid structures (example, thymus,Waldeyer's ring) on both sides of the diaphragm with optional localised extranodal site (IIIE) or spleen (IIIS); stage IV-Diffuse or disseminated extralymphatic organ involvement.
Prognostic Index Score | Baseline
  Prognostic index will be summarized using descriptive statistics. For each prognostic factor, 0-3 points are given to each patient and points are summed up to a maximum of 11. Participants with 0-3 points are classified as low risk (44% of participants, median overall survival [OS] not reached). Participants with 4-5 points are classified as intermediate risk (35%, median OS 51 months), and patients with 6-11 points as high risk (21%, median OS 29 months).
Demographic Characteristic of Participants in Prospective Group: Gender | Baseline
  Categorical variable (gender) will be summarized using a frequency distribution with the number and percentage of participants in each category.
Treatment pattern of BTZ-treated MCL participants: Route of Administration | Up to Follow-up (approximately 22 months)
  Primary MCL therapy with Velcade (BTZ) prior MCL treatment, combined MCL treatment and subsequent MCL treatment to extract the information on route of administration (subcutaneous [SC] or intravenous [IV]) to see if there's any outstanding factor that impacts BTZ's dose/frequency and identify the most popular usage of BTZ.
Treatment Pattern of Bortezomib (BTZ) Treated MCL participants: Dose | Up to Follow-up (approximately 22 months)
  The cumulated dose will be summarized using descriptive statistics.
Treatment Pattern of Bortezomib (BTZ) Treated MCL Participants: Frequency | Up to Follow-up (approximately 22 months)
  The frequency of BTZ will be summarized using a frequency distribution with the number and percentage of participants in each category.
Treatment Pattern of Bortezomib (BTZ) Treated MCL Participants: Reason of BTZ Initiation/Discontinuation/Dose Adjustment | Up to Follow-up (approximately 22 months)
  The reason of BTZ initiation/discontinuation/dose adjustment will be described with respective number of occurrence.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 22 months
  ORR is defined as the sum of complete response [CR] rate (CR+ unconfirmed complete remission [CRu]) + Partial remission [PR] rate as per International Working Group (IWG 2007) criteria. These response criteria are based on the reduction in the size of the enlarged lymph node as measured by computerized tomography (CT) scan and the extent of bone marrow involvement that is determined by bone marrow aspirate and biopsy. Complete response [CR] defined as disappearance of all evidence of disease; CRu satisfies CR criteria, however any residual lymph node mass greater than (>)1.5 centimeter (cm) in longest transverse dimension or extranodal site of disease (irrespective of size) must have regressed by more than 75% of the product of the longest perpendicular dimensions compared to the pretreatment baseline. PR defined as at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses.
Complete Response [CR] Rate (CR+ Unconfirmed Complete Remission CRu) | Approximately 22 months
  The percentage of participants with CR and CRu in all participants whose treatment response data are available.
Partial Remission (PR) Rate | Approximately 22 months
  The percentage of participants with PR in all participants whose treatment response data are available.
Time to Response (TTR) | Approximately 22 months
  Interval between start of treatment to the first day when CR/CRu or PR was observed.
Duration of Response (DOR) | Approximately 22 months
  Interval from the date the response was documented to the first day that Progressive Disease (PD) was observed in participants with CR/CRu or PR. PD defined as any new lesions or increase by greater than or equal to (>=) 50% of previously involved sites from nadir.
Progressive-Free Survival (PFS) | Approximately 22 months
  Interval between start of treatment to first day when death or PD was observed. PD defined as any new lesions or increase by >= 50% of previously involved sites from nadir.
Overall survival (OS) | Approximately 22 months
  Interval from the day of the start of the treatment to death, or the last date when the participant was identified to be alive whichever is late.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (9):
- China (9):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Nanfang Hospital, Guangzhou
  - Jiangsu Province Hospital, Nanjing
  - Ruijin Hospital, Shanghai Jiao Tong University, Shanghai
  - Huashan Hospital Fudan University, Shanghai
  - Blood Disease Hospital of Chinese Academy of Medical Sciences, Tianjin